CLINICAL TRIAL: NCT02683785
Title: A Multi-centre Phase IIa Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of GSK3196165 in Subjects With Inflammatory Hand Osteoarthritis
Brief Title: A Study to Investigate the Efficacy and Safety of GSK3196165 in Inflammatory Hand Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 204851; 2015-003089-96 (EudraCT Number)
Record Dates: First submitted 2016-01-21; First posted 2016-02-17 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis
Keywords: Pain intensity; Hand Osteoarthritis; GSK3196165; AUSCAN; GM-CSF; Numerical Rating Scale
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Otilimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK3196165 (Experimental): Subjects will receive a total of 8 doses of GSK3196165 over a 12-week treatment period.
  Interventions: Drug: GSK3196165
- Placebo (Placebo Comparator): Subjects will receive a total of 8 doses of placebo over a 12-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3196165 — GSK3196165 will be supplied as a liquid and will be administered as a subcutaneous injection. The drug will be administered weekly for 5 injections, then every other week for 3 further injections.
  Arms: GSK3196165
Drug: Placebo — Matching placebo will be administered as above.
  Arms: Placebo

SUMMARY:
This is a randomized, Phase IIa, multicentre, double-blind, placebo-controlled parallel group study with the primary objective to assess the efficacy potential of GSK3196165 on pain, in subjects with active inflammatory hand osteoarthritis (HOA).

Approximately 40 subjects will be enrolled into the study, following a screening period of up to 4 weeks. The total treatment period will be 12 weeks, with the follow up period completing at Week 22. At least 40 subjects will be randomized across the two treatment arms, to either placebo or GSK3196165 in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years at the time of signing informed consent.
* Meets American College of Rheumatology (ACR) classification of osteoarthritis (OA) and have not responded to analgesics (level 1 and 2) or to non-steroidal anti-inflammatory drugs (NSAIDs) for at least 10 days in the past 3 months.
* Active disease at screening and randomization with at least two swollen and tender proximal interphalangeal (PIP) and/or distal interphalangeal (DIP) joints in the affected hand.
* Signs of inflammation such as synovitis in the MRI scan of the affected hand.
* Must have a subject's self assessment of 24-hour average hand pain intensity at baseline of at least '5' on an 11-point Numerical Rating Scale (NRS, 0-10).
* Weight >=45 kilogram (kg).
* Male or female subjects are eligible to participate so long as they meet and agree to abide by the contraceptive criteria.
* Diffusing capacity of the lung for carbon monoxide (DLCO) >=70% predicted; forced expiratory volume in 1 second (FEV1) >=80% predicted.
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

* Pregnant or lactating women.
* History of any clinically significant inflammatory disease other than inflammatory HOA, especially, but not limited to, rheumatoid arthritis or spondylarthropathies.
* Diagnosis of rheumatoid arthritis, fibromyalgia, gout, calcium pyrophosphate deposition disease (CPPD), pseudogout, hemochromatosis or other inflammatory rheumatological or autoimmune disorders.
* Clinical suspicion of, or previous investigation for CPPD or pseudogout, or history of chondrocalcinosis.
* Any injury, medical or surgical procedure to the affected joint(s) that may interfere with evaluation of the target HOA joint(s).
* History of infected joint prosthesis at any time, with the prosthesis still in situ. History of leg ulcers, catheters, chronic sinusitis or recurrent chest or urinary tract infections.
* Any surgical procedure, including bone or joint surgery/synovectomy within 12 weeks prior to Day 1 or any planned surgery within the duration of the study or follow-up period.
* History of any respiratory disease which (in the opinion of the investigator) would compromise subject safety or the ability of the subject to complete the study (e.g. significant interstitial lung disease, such as pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), moderate-severe asthma, bronchiectasis, previous pulmonary alveolar proteinosis [PAP]).
* Clinically-significant or unstable (in the opinion of the investigator) persistent cough or dyspnea that is unexplained.
* Significant unstable or uncontrolled acute or chronic disease which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* A history of malignancy.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* Current/previous Hepatitis B virus (HBV), Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) 1 or 2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Duncansville, Pennsylvania
- Germany (3):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
- Netherlands (3):
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Nowa Sól
  - GSK Investigational Site, Warsaw
- United Kingdom (4):
  - GSK Investigational Site, Canterbury, Kent
  - GSK Investigational Site, Derby
  - GSK Investigational Site, North Shields
  - GSK Investigational Site, York

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20746

REFERENCES:
- [Background] Georg Schett, Chris Bainbridge, Mario Berkowitz, Katherine Davy, Sofia Fernandes, Eduard Griep, Stephen Harrison, James Lloyd-Hughes, Alexandra Morgan-Roberts, Mark Layton, Nonna Anna Nowak, Jatin Patel, Jürgen Rech, Sarah Watts, Paul P. Tak. A Phase IIa, randomised study of the safety, pharmacokinetics, pharmacodynamics and clinical activity of the anti-GM-CSF antibody GSK3196165 in patients with hand osteoarthritis. Lancet Rheumatol. 2020; DOI: 10.1016/S2665-9913(20)30171-5
- [Derived] Schett G, Bainbridge C, Berkowitz M, Davy K, Fernandes S, Griep E, Harrison S, Gupta A, Lloyd-Hughes J, Roberts A, Layton M, Nowak NA, Patel J, Rech J, Smith JE, Watts S, Tak PP. Anti-granulocyte-macrophage colony-stimulating factor antibody otilimab in patients with hand osteoarthritis: a phase 2a randomised trial. Lancet Rheumatol. 2020 Oct;2(10):e623-e632. doi: 10.1016/S2665-9913(20)30171-5. Epub 2020 Sep 23. PMID 38273625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, double-blind, placebo-controlled study to investigate the efficacy and safety of GSK3196165 in participants with inflammatory hand osteoarthritis. The study was conducted in five countries in Poland, United Kingdom, Netherlands, Germany and United States.
Pre-assignment Details: A total 121 participants were screened of which 77 were screen failures and 44 participants were enrolled in the study.
Groups:
- Placebo: Participants randomized to Placebo group received total of 8 subcutaneous injections of placebo over a 12-week treatment period. Participants were administered loading doses on Days 1, 8, 15, 22 and 29 which was followed by 3 doses every other week (Days 43, 57, 71).
- GSK3196165 180mg: Participants randomized to GSK3196165 group received total of 8 doses of GSK3196165 over a 12-week treatment period. Participants were administered loading doses on Days 1, 8, 15, 22 and 29 which was followed by 3 doses every other week (Days 43, 57, 71).
Period: Overall Study
Arm/Group | Placebo | GSK3196165 180mg
Started | 22 | 22
Completed | 21 | 18
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3196165 180mg | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (6.80) | 60.9 (6.25) | 58.8 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White /Caucasian/European | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Average Hand Pain Intensity, Averaged Over the 7 Days Prior to Week 6
Description: Participants were required to complete a daily pain NRS based on their 24-hour average hand pain intensity with the anchors "0" (no pain) and "10" (worst imaginable pain), which was averaged over the 7 days prior to assessment visit. The 7 day average score was calculated as sum of daily 24 hours average hand pain NRS scores in the 7 days prior to assessment visit, divided by number of entries recorded in those 7 days. Baseline visit was at Day 1 and Baseline value was defined as the average of the 7 days prior to baseline visit (Day 1 pre-dose). Change from Baseline is equal to post-dose visit value minus Baseline value. Intent-To-Treat Population comprised of all randomized participants who received at least one dose of study treatment (GSK3196165 or placebo).
Time Frame: Baseline (Day 1 Pre-dose) and Week 6
Population: Intent To Treat Population. Only non-missing data is included MMRM model.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 21 | 20
Scores on scale | -1.34 (0.325) | -1.70 (0.334)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.442, Mixed Model Repeated Measures Analysis — MMRM model with fixed effects of Baseline Value,Treatment Group,Visit and Treatment Group by Visit Interaction was used. Unstructured covariance structure was used.p-value corresponds to the difference over placebo measure and confidence interval; Mean Difference (Net) = -0.36, 95% CI 2-sided [-1.31 to 0.58] — Difference from placebo for Week 6 is presented

2. Secondary Outcome: Change From Baseline in 24 Hours Average Hand Pain Intensity Averaged Over the 7 Days Prior to Each Visit
Description: Participants were required to complete a daily pain NRS based on their 24-hour average hand pain intensity with the anchors "0" (no pain) and "10" (worst imaginable pain), which was averaged over the 7 days prior to assessment visit. The 7 day average score is calculated by sum of daily 24 hours average hand pain NRS scores in the 7 days prior to assessment visit, divided by number of entries recorded in those 7 days. Baseline visit was at Day 1 and Baseline value was defined as the average of the 7 days prior to baseline visit (Day 1 pre-dose). Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose Day 1), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Intent To Treat Population. n=X in category titles represents the number of participants with non-missing data at the specified time-point. Only non-missing data is included in the MMRM model.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Week 1, n=22, 20: number analyzed (Participants) | 22 | 20
  Week 1, n=22, 20 | -0.13 (0.152) | -0.59 (0.160)
  Week 2, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 2, n=21, 20 | -0.48 (0.230) | -0.86 (0.239)
  Week 3, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 3, n=21, 20 | -0.74 (0.279) | -1.24 (0.289)
  Week 4, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 4, n=21, 20 | -0.91 (0.291) | -1.65 (0.301)
  Week 6, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 6, n=21, 20 | -1.34 (0.325) | -1.70 (0.334)
  Week 8, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 8, n=20, 19 | -1.27 (0.382) | -2.10 (0.393)
  Week 10, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 10, n=20, 19 | -1.18 (0.376) | -2.09 (0.389)
  Week 12, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 12, n=19, 18 | -1.35 (0.402) | -2.24 (0.416)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.046, Mixed Model Repeated Measures Analysis — MMRM model with fixed effects of Baseline Value, Treatment Group, Visit and Treatment Group by Visit Interaction was used. Unstructured covariance structure was used. p-value corresponds to the difference over placebo measure and confidence interval; Mean Difference (Net) = -0.46, 95% CI 2-sided [-0.90 to -0.01] — Difference from placebo for Week 1 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.257, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.38, 95% CI 2-sided [-1.05 to 0.29] — Difference from placebo for Week 2 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.220, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.50, 95% CI 2-sided [-1.31 to 0.31] — Difference from placebo for Week 3 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.085, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.74, 95% CI 2-sided [-1.59 to 0.11] — Difference from placebo for Week 4 is presented
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.442, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.36, 95% CI 2-sided [-1.31 to 0.58] — Difference from placebo for Week 6 is presented
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.139, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.93 to 0.28] — Difference from placebo for Week 8 is presented
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.103, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.90, 95% CI 2-sided [-2.00 to 0.19] — Difference from placebo for Week 10 is presented
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.132, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.89, 95% CI 2-sided [-2.06 to 0.28] — Difference from placebo for Week 12 is presented

3. Secondary Outcome: Change From Baseline of Worst Hand Pain Intensity Over 24 Hours Averaged Over the 7 Days Prior to Each Visit
Description: Participants were required to complete a daily pain NRS based on their 24-hour worst hand pain intensity with the anchors "0" (no pain) and "10" (worst imaginable pain), which was averaged over the 7 days prior to assessment visit. The score is calculated as sum of daily 24 hours worst hand pain NRS scores in the 7 days prior to assessment visit, divided by number of entries recorded in those 7 days. Baseline visit was at Day 1 and Baseline value was defined as the average of the 7 days prior to baseline visit (Day 1 pre-dose). Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose Day 1), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Intent-to-Treat Population. n=X in category titles represents the number of participants with non-missing data at the specified time-point. Only non-missing data is included in the MMRM model.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Week 1, n=22, 20: number analyzed (Participants) | 22 | 20
  Week 1, n=22, 20 | 0.01 (0.174) | -0.45 (0.183)
  Week 2, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 2, n=21, 20 | -0.42 (0.235) | -0.69 (0.245)
  Week 3, n=21, 20: number analyzed (Participants) | 21 | 20
  Week 3, n=21, 20 | -0.63 (0.269) | -1.23 (0.278)
  Week 4, n= 21, 20: number analyzed (Participants) | 21 | 20
  Week 4, n= 21, 20 | -0.72 (0.289) | -1.51 (0.299)
  Week 6, n= 21, 20: number analyzed (Participants) | 21 | 20
  Week 6, n= 21, 20 | -1.30 (0.328) | -1.63 (0.337)
  Week 8, n= 20, 19: number analyzed (Participants) | 20 | 19
  Week 8, n= 20, 19 | -1.18 (0.394) | -2.11 (0.406)
  Week 10, n= 20, 19: number analyzed (Participants) | 20 | 19
  Week 10, n= 20, 19 | -1.15 (0.394) | -2.13 (0.407)
  Week 12, n= 19, 18: number analyzed (Participants) | 19 | 18
  Week 12, n= 19, 18 | -1.32 (0.415) | -2.34 (0.430)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.082, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.97 to 0.06] — Difference from placebo for Week 1 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.426, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.96 to 0.41] — Difference from placebo for Week 2 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.129, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.60, 95% CI 2-sided [-1.38 to 0.18] — Difference from placebo for Week 3 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.067, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.78, 95% CI 2-sided [-1.63 to 0.06] — Difference from placebo for Week 4 is presented
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.494, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-1.28 to 0.63] — Difference from placebo for Week 6 is presented
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.107, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.94, 95% CI 2-sided [-2.08 to 0.21] — Difference from placebo for Week 8 is presented
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.092, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.98, 95% CI 2-sided [-2.13 to 0.17] — Difference from placebo for Week 10 is presented
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.098, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.01, 95% CI 2-sided [-2.22 to 0.20] — Difference from placebo for Week 12 is presented

4. Secondary Outcome: Percentage of Participants Achieving a 30 Percentage Reduction From Baseline in 24 Hours Average Hand Pain Intensity at Each Visit
Description: Participants were required to complete average pain NRS daily and rate the average hand pain over last 24 hours on a scale of 0 (no pain) to 10 (worst imaginable pain). The percentage of participants who achieved at least 30 percentage reduction from Baseline in the 24-hours average hand pain intensity as measured by daily NRS and averaged over 7 days prior to each visit is reported.
Time Frame: Baseline (Pre-dose, Day 1), Weeks 1, 2, 3, 4, 6, 8, 10, 12 and follow up (Week 22)
Population: Intent-to-Treat Population. Participants with missing data at a particular visit had been assumed to be non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Percentage of participants
  Week 1 | 0 | 9
  Week 2 | 0 | 18
  Week 3 | 5 | 23
  Week 4 | 14 | 41
  Week 6 | 23 | 45
  Week 8 | 18 | 50
  Week 10 | 18 | 50
  Week 12 | 23 | 45
  Follow up (Week 22) | 23 | 27

5. Secondary Outcome: Percentage of Participants Achieving a 50 Percentage Reduction From Baseline in 24 Hours Average Hand Pain Intensity at Each Visit
Description: Participants were required to complete average pain NRS daily and rate the average hand pain over last 24 hours on a scale of 0 (no pain) to 10 (worst imaginable pain). The percentage of participants who achieved at least 50 percentage reduction from Baseline in the 24-hours average hand pain intensity as measured by daily NRS and averaged over 7 days prior to each visit is presented.
Time Frame: Baseline (Pre-dose, Day 1), Weeks 1, 2, 3, 4, 6, 8, 10, 12 and follow up (Week 22)
Population: Intent-to-Treat Population. Participants with missing data at a particular visit had been assumed to be non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Percentage of participants
  Week 1 | 0 | 0
  Week 2 | 0 | 9
  Week 3 | 0 | 18
  Week 4 | 0 | 23
  Week 6 | 14 | 27
  Week 8 | 14 | 41
  Week 10 | 9 | 36
  Week 12 | 14 | 41
  Follow up (Week 22) | 9 | 23

6. Secondary Outcome: Percentage of Participants Achieving a 30 Percentage Reduction From Baseline in 24 Hours Worst Hand Pain Intensity at Each Visit
Description: Participants were required to complete worst pain NRS daily and rate the hand pain at its worst over last 24 hours on a scale of 0 (no pain) to 10 (worst imaginable pain). The percentage of participants achieving at least 30 percentage reduction from Baseline in the 24-hours worst hand pain intensity as measured by daily NRS and averaged over 7 days prior to each visit is presented.
Time Frame: Baseline (Pre-dose, Day 1), Weeks 1, 2, 3, 4, 6, 8, 10, 12 and follow up (Week 22)
Population: Intent-to-Treat Population. Participants with missing data at a particular visit had been assumed to be non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Percentage of participants
  Week 1 | 0 | 9
  Week 2 | 0 | 18
  Week 3 | 0 | 23
  Week 4 | 0 | 32
  Week 6 | 9 | 36
  Week 8 | 9 | 45
  Week 10 | 14 | 45
  Week 12 | 14 | 45
  Follow up (Week 22) | 14 | 32

7. Secondary Outcome: Percentage of Participants Achieving a 50 Percentage Reduction From Baseline in 24 Hours Worst Hand Pain Intensity at Each Visit
Description: Participants were required to complete worst pain NRS daily and rate the hand pain at its worst over last 24 hours on a scale of 0 (no pain) to 10 (worst imaginable pain). The percentage of participants achieving at least 50 percentage reduction from Baseline in the 24-hours worst hand pain intensity as measured by daily NRS and averaged over 7 days prior to each visit is presented.
Time Frame: Baseline (Pre-dose, Day 1), Weeks 1, 2, 3, 4, 6, 8, 10, 12 and follow up (Week 22)
Population: Intent-to-Treat Population. Participants with missing data at a particular visit had been assumed to be non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Percentage of participants
  Week 1 | 0 | 0
  Week 2 | 0 | 5
  Week 3 | 0 | 14
  Week 4 | 0 | 18
  Week 6 | 5 | 18
  Week 8 | 5 | 32
  Week 10 | 5 | 27
  Week 12 | 9 | 36
  Follow up (Week 22) | 5 | 23

8. Secondary Outcome: Change From Baseline in Australian Canadian Hand Osteoarthritis Index (AUSCAN) 3.1 NRS Scores at Each Visit.
Description: The AUSCAN Index is a self-administered questionnaire consisting of a 15-item scale which measures pain (5 items), stiffness (1 item) and degree of disability/physical function (9 items) during the preceding 48 hours. All items are rated on NRS scale with anchors "0" (none) to "10" (extreme). The scores for the pain and physical function components were calculated as simple summation of the item scores relating to that domain, so the Pain component ranges from 0 (i.e. all pain item scores are scored 0 [none]) to 50 (i.e. all pain item scores are scored 10 [extreme]), and the Physical Function component ranges from 0 (i.e. all physical function item scores are scored 0 [none]) to 90 (i.e. all physical function item scores are scored 10 [extreme]). The total AUSCAN score was calculated as simple summation of the 15 item scores and therefore ranges from 0 to 150. Baseline is defined as Day 1 pre-dose value. Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 Pre-dose), Weeks 1, 2, 4, 6, 8, 10, and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Pain, Week 1, n=22, 20: number analyzed (Participants) | 22 | 20
  Pain, Week 1, n=22, 20 | 0.8 (0.98) | -1.9 (1.03)
  Pain, Week 2, n=21, 21: number analyzed (Participants) | 21 | 21
  Pain, Week 2, n=21, 21 | -1.8 (1.27) | -3.7 (1.28)
  Pain, Week 4, n=22, 21: number analyzed (Participants) | 22 | 21
  Pain, Week 4, n=22, 21 | -3.5 (1.61) | -7.2 (1.64)
  Pain, Week 6, n=22, 21: number analyzed (Participants) | 22 | 21
  Pain, Week 6, n=22, 21 | -6.6 (1.72) | -7.6 (1.76)
  Pain, Week 8, n=20, 20: number analyzed (Participants) | 20 | 20
  Pain, Week 8, n=20, 20 | -4.9 (1.93) | -8.7 (1.97)
  Pain, Week 10, n=20, 20: number analyzed (Participants) | 20 | 20
  Pain, Week 10, n=20, 20 | -5.3 (1.82) | -10.9 (1.87)
  Pain, Week 12, n=21, 19: number analyzed (Participants) | 21 | 19
  Pain, Week 12, n=21, 19 | -4.6 (1.84) | -9.3 (1.91)
  Stiffness, Week 1, n= 22, 20: number analyzed (Participants) | 22 | 20
  Stiffness, Week 1, n= 22, 20 | -0.4 (0.29) | -0.6 (0.31)
  Stiffness, Week 2, n= 21, 21: number analyzed (Participants) | 21 | 21
  Stiffness, Week 2, n= 21, 21 | -0.8 (0.33) | -1.1 (0.33)
  Stiffness, Week 4, n= 22, 21: number analyzed (Participants) | 22 | 21
  Stiffness, Week 4, n= 22, 21 | -1.2 (0.41) | -1.8 (0.42)
  Stiffness, Week 6, n= 22, 21: number analyzed (Participants) | 22 | 21
  Stiffness, Week 6, n= 22, 21 | -1.4 (0.39) | -1.6 (0.40)
  Stiffness, Week 8, n= 20, 20: number analyzed (Participants) | 20 | 20
  Stiffness, Week 8, n= 20, 20 | -1.2 (0.41) | -1.9 (0.42)
  Stiffness, Week 10, n= 20, 20: number analyzed (Participants) | 20 | 20
  Stiffness, Week 10, n= 20, 20 | -1.6 (0.44) | -2.2 (0.45)
  Stiffness, Week 12, n= 21, 19: number analyzed (Participants) | 21 | 19
  Stiffness, Week 12, n= 21, 19 | -1.5 (0.45) | -2.2 (0.47)
  Physical function, Week 1, n=22, 20: number analyzed (Participants) | 22 | 20
  Physical function, Week 1, n=22, 20 | -0.7 (2.08) | -3.6 (2.16)
  Physical function, Week 2, n=21,21: number analyzed (Participants) | 21 | 21
  Physical function, Week 2, n=21,21 | -2.8 (2.35) | -5.7 (2.37)
  Physical function, Week 4, n=22, 21: number analyzed (Participants) | 22 | 21
  Physical function, Week 4, n=22, 21 | -6.4 (3.01) | -11.3 (3.07)
  Physical function, Week 6, n=22, 21: number analyzed (Participants) | 22 | 21
  Physical function, Week 6, n=22, 21 | -9.1 (3.25) | -11.8 (3.32)
  Physical function, Week 8, n=20, 20: number analyzed (Participants) | 20 | 20
  Physical function, Week 8, n=20, 20 | -8.3 (3.57) | -13.2 (3.64)
  Physical function, Week 10, n=20, 20: number analyzed (Participants) | 20 | 20
  Physical function, Week 10, n=20, 20 | -9.0 (3.82) | -15.2 (3.92)
  Physical function, Week 12, n=21, 19: number analyzed (Participants) | 21 | 19
  Physical function, Week 12, n=21, 19 | -7.2 (3.74) | -15.4 (3.87)
  Total, Week 1, n= 22, 20: number analyzed (Participants) | 22 | 20
  Total, Week 1, n= 22, 20 | -0.5 (3.07) | -6.0 (3.20)
  Total, Week 2, n= 21, 21: number analyzed (Participants) | 21 | 21
  Total, Week 2, n= 21, 21 | -5.7 (3.66) | -10.4 (3.70)
  Total, Week 4, n= 22, 21: number analyzed (Participants) | 22 | 21
  Total, Week 4, n= 22, 21 | -11.4 (4.72) | -20.1 (4.83)
  Total, Week 6, n= 22, 21: number analyzed (Participants) | 22 | 21
  Total, Week 6, n= 22, 21 | -17.3 (5.17) | -20.7 (5.28)
  Total, Week 8, n= 20, 20: number analyzed (Participants) | 20 | 20
  Total, Week 8, n= 20, 20 | -14.6 (5.70) | -23.6 (5.81)
  Total, Week 10, n= 20, 20: number analyzed (Participants) | 20 | 20
  Total, Week 10, n= 20, 20 | -16.1 (5.88) | -28.2 (6.04)
  Total, Week 12, n= 21, 19: number analyzed (Participants) | 21 | 19
  Total, Week 12, n= 21, 19 | -13.5 (5.92) | -26.7 (6.12)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.061, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.8, 95% CI 2-sided [-5.6 to 0.1] — For Pain component, Week 1
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.282, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.0, 95% CI 2-sided [-5.6 to 1.7] — For Pain component, Week 2
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.113, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.7, 95% CI 2-sided [-8.4 to 0.9] — For Pain component Week 4
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.695, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.0, 95% CI 2-sided [-5.9 to 4.0] — For Pain component, Week 6
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.176, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.8, 95% CI 2-sided [-9.4 to 1.8] — For Pain component, Week 8
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.041, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -5.5, 95% CI 2-sided [-10.8 to -0.2] — For Pain component, Week 10
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.082, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.7, 95% CI 2-sided [-10.1 to 0.6] — For Pain component, Week 12
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.587, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.1 to 0.6] — For Stiffness component, Week 1
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.457, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.3 to 0.6] — For Stiffness component, Week 2
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.298, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.8 to 0.6] — For Stiffness component, Week 4
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.726, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.3 to 0.9] — For Stiffness component, Week 6
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.213, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.9 to 0.4] — For Stiffness component, Week 8
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.331, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.9 to 0.7] — For Stiffness component, Week 10
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.248, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.1 to 0.6] — For Stiffness component, Week 12
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.350, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.9, 95% CI 2-sided [-9.0 to 3.3] — For Physical Function component, Week 1
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.383, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.0, 95% CI 2-sided [-9.8 to 3.8] — For Physical Function component, Week 2
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.271, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.8, 95% CI 2-sided [-13.5 to 3.9] — For Physical Function component, Week 4
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.565, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.7, 95% CI 2-sided [-12.1 to 6.7] — For Physical Function component, Week 6
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.343, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.9, 95% CI 2-sided [-15.2 to 5.4] — For Physical Function component, Week 8
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.266, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -6.2, 95% CI 2-sided [-17.3 to 4.9] — For Physical Function component, Week 10
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.136, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -8.2, 95% CI 2-sided [-19.1 to 2.7] — For Physical Function component, Week 12
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.230, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -5.5, 95% CI 2-sided [-14.5 to 3.6] — For Total of all component scores, Week 1
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.381, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.6, 95% CI 2-sided [-15.2 to 5.9] — For Total of all component scores, Week 2
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.207, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -8.7, 95% CI 2-sided [-22.4 to 5.0] — For Total of all component scores, Week 4
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.648, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.4, 95% CI 2-sided [-18.4 to 11.6] — For Total of all component scores, Week 6
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.278, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -9.0, 95% CI 2-sided [-25.4 to 7.5] — For Total of all component scores, Week 8
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.160, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -12.1, 95% CI 2-sided [-29.1 to 5.0] — For Total of all component scores, Week 10
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.127, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -13.3, 95% CI 2-sided [-30.5 to 3.9] — For Total of all component scores, Week 12

9. Secondary Outcome: Change From Baseline in Number of Soft Tissue Swollen Hand Joints at Each Visit
Description: Swollen Hand Joint Count was measured by the total number of soft tissue swollen hand joints out of a possible 30 joints: 8 distal interphalangeal, 8 proximal interphalangeal, 2 interphalangeal joints, 10 metacarpophalangeal joints, 2 carpometacarpal joint across both hands. In case of missing observations for soft tissue swollen hand joints then the remaining observations were assessed and weighted by dividing the number presented by the number of non-missing, and by multiplying by 30 for the joint count. Baseline is defined as Day 1 pre-dose value. Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 Pre-dose), Weeks 1, 2, 4, 6, 8, 10, and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Swollen joints
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Swollen joints
  Week 1, n = 22, 21: number analyzed (Participants) | 22 | 21
  Week 1, n = 22, 21 | -0.3 (0.64) | -0.3 (0.66)
  Week 2, n = 21, 21: number analyzed (Participants) | 21 | 21
  Week 2, n = 21, 21 | -1.6 (0.85) | -1.2 (0.86)
  Week 4, n = 22, 21: number analyzed (Participants) | 22 | 21
  Week 4, n = 22, 21 | -1.6 (0.76) | -2.1 (0.78)
  Week 6, n = 22, 21: number analyzed (Participants) | 22 | 21
  Week 6, n = 22, 21 | -3.7 (0.83) | -2.3 (0.85)
  Week 8, n = 20, 20: number analyzed (Participants) | 20 | 20
  Week 8, n = 20, 20 | -3.0 (0.92) | -2.8 (0.94)
  Week 10, n = 20, 20: number analyzed (Participants) | 20 | 20
  Week 10, n = 20, 20 | -2.6 (1.08) | -2.9 (1.10)
  Week 12, n = 21, 19: number analyzed (Participants) | 21 | 19
  Week 12, n = 21, 19 | -2.9 (0.91) | -3.1 (0.93)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.957, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.9 to 1.8] — Difference from placebo for Week 1 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.775, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.1 to 2.8] — Difference from placebo for Week 2 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.624, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.7 to 1.7] — Difference from placebo for Week 4 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.243, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 1.4, 95% CI 2-sided [-1.0 to 3.8] — Difference from placebo for Week 6 is presented
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.875, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.2, 95% CI 2-sided [-2.5 to 2.9] — Difference from placebo for Week 8 is presented
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.848, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.3, 95% CI 2-sided [-3.4 to 2.8] — Difference from placebo for Week 10 is presented
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.883, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-2.8 to 2.4] — Difference from placebo for Week 12 is presented

10. Secondary Outcome: Change From Baseline in Number of Tender Hand Joints at Each Visit
Description: Tender Hand Joint Count was measured by the total number of tender joints out of a possible 30 joints: 8 distal interphalangeal, 8 proximal interphalangeal, 2 interphalangeal joints, 10 metacarpophalangeal joints, 2 carpometacarpal joints across both hands. A joint was considered tender if it was scored >0 on the tender joint severity scale. Joints were rated 0=no pain/tenderness, 1=mild pain, 2=moderate pain and 3=severe pain. Baseline is defined as Day 1 pre-dose value. Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Intent-to-Treat Population. n=X in category titles represents the number of participants with non-missing data at the specified time-point. Only non-missing data was included in the MMRM model.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Week 1, n= 22, 21: number analyzed (Participants) | 22 | 21
  Week 1, n= 22, 21 | -0.6 (1.10) | -1.8 (1.13)
  Week 2, n= 21, 21: number analyzed (Participants) | 21 | 21
  Week 2, n= 21, 21 | -1.7 (1.15) | -2.1 (1.17)
  Week 4, n= 22, 21: number analyzed (Participants) | 22 | 21
  Week 4, n= 22, 21 | -1.1 (1.33) | -3.0 (1.36)
  Week 6, n= 22, 21: number analyzed (Participants) | 22 | 21
  Week 6, n= 22, 21 | -3.7 (1.27) | -4.2 (1.30)
  Week 8, n= 20, 20: number analyzed (Participants) | 20 | 20
  Week 8, n= 20, 20 | -2.4 (1.36) | -3.9 (1.39)
  Week 10, n= 20, 20: number analyzed (Participants) | 20 | 20
  Week 10, n= 20, 20 | -3.7 (1.45) | -4.4 (1.48)
  Week 12, n= 21, 19: number analyzed (Participants) | 21 | 19
  Week 12, n= 21, 19 | -3.5 (1.46) | -4.0 (1.51)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.463, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.2, 95% CI 2-sided [-4.4 to 2.0] — Difference from placebo for Week 1 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.809, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-3.7 to 2.9] — Difference from placebo for Week 2 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.324, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.9, 95% CI 2-sided [-5.8 to 2.0] — Difference from placebo for Week 4 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.783, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-4.2 to 3.2] — Difference from placebo for Week 6 is presented
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.464, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.4, 95% CI 2-sided [-5.4 to 2.5] — Difference from placebo for Week 8 is presented
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.736, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.9 to 3.5] — Difference from placebo for Week 10 is presented
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.806, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-4.8 to 3.7] — Difference from placebo for Week 12 is presented

11. Secondary Outcome: Change From Baseline in Physician Global Assessment (PhGA) of Disease Activity
Description: Physicians were required to complete the global assessment of disease activity using single PhGA item with a NRS ranging from 0 (none) to 10 (extremely active). Baseline was defined as Day 1 pre-dose value. Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 Pre-dose), Weeks 2, 4, 8, and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Week 2, n= 19, 14: number analyzed (Participants) | 19 | 14
  Week 2, n= 19, 14 | -1.8 (0.39) | -1.5 (0.45)
  Week 4, n= 20, 15: number analyzed (Participants) | 20 | 15
  Week 4, n= 20, 15 | -2.1 (0.44) | -2.6 (0.50)
  Week 8, n= 17, 15: number analyzed (Participants) | 17 | 15
  Week 8, n= 17, 15 | -2.2 (0.52) | -3.4 (0.57)
  Week 12, n= 18, 14: number analyzed (Participants) | 18 | 14
  Week 12, n= 18, 14 | -2.7 (0.56) | -3.0 (0.63)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.586, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.9 to 1.6] — Difference from placebo for Week 2 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.416, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.9 to 0.8] — Difference from placebo for Week 4 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.120, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.8 to 0.3] — Difference from placebo for Week 8 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.687, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.1 to 1.4] — Difference from placebo for Week 12 is presented

12. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) of Disease Activity
Description: Participants were required to complete the global assessment of disease activity using single PtGA item with an NRS ranging from 0 (very well) to 10 (very poor). Baseline was defined as Day 1 pre-dose value. Change from Baseline is equal to post-dose visit value minus Baseline value.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Scores on scale
  Week 2, n= 20, 21: number analyzed (Participants) | 20 | 21
  Week 2, n= 20, 21 | -0.4 (0.36) | -0.6 (0.35)
  Week 4, n= 21, 21: number analyzed (Participants) | 21 | 21
  Week 4, n= 21, 21 | -0.6 (0.42) | -1.3 (0.42)
  Week 8, n= 19, 20: number analyzed (Participants) | 19 | 20
  Week 8, n= 19, 20 | -0.9 (0.47) | -1.8 (0.46)
  Week 12, n= 20, 19: number analyzed (Participants) | 20 | 19
  Week 12, n= 20, 19 | -0.7 (0.46) | -1.8 (0.46)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.651, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.3 to 0.8] — Difference from placebo for Week 2 is presented
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.271, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.9 to 0.5] — Difference from placebo for Week 4 is presented
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.186, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.2 to 0.4] — Difference from placebo for Week 8 is presented
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180mg; Test type: Other; p = 0.109, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.4 to 0.2] — Difference from placebo for Week 12 is presented

13. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or events associated with liver injury and impaired liver function were categorized as SAE. All participants who received at least one dose of study treatment (GSK3196165 or placebo) were included in Safety Population.
Time Frame: Up to Week 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Participants
  Any AE | 11 | 13
  Any SAE | 1 | 2

14. Secondary Outcome: Number of Participants With Infections
Description: Adverse events of special interest (AESI) included serious infections like serious respiratory infections and tuberculosis and other opportunistic infections. Number of participants with infections has been reported.
Time Frame: Up to Week 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Participants
  Serious Infections | 0 | 0
  Opportunistic Infections | 0 | 0

15. Secondary Outcome: Number of Participants With Pulmonary Events
Description: Pulmonary events like pulmonary alveolar proteinosis (PAP), persistent (for 3 consecutive weeks) reduction in diffusing capacity of the lungs for carbon monoxide (DLCO) > 15 percentage, persistent (for 3 consecutive weeks) cough and/or dyspnea and non- life threatening pulmonary changes related to surfactant accumulation is presented.
Time Frame: Up to Week 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Participants
  Persistent dyspnea | 0 | 0
  Persistent decrease in DLCO | 0 | 0
  Persistent Cough | 0 | 0
  Abnormal Lung Auscultation | 0 | 0
  PAP | 0 | 0

16. Secondary Outcome: Number of Participants With Anti-GSK3196165 Binding Antibodies
Description: Serum samples were collected at indicated time points for anti-drug antibody (ADA) measurements. Anti-GSK3196165 binding antibody detection assay using tiered testing schema: screening, confirmation and titration steps was used for immunogenicity analysis. Samples taken after dosing with GSK3196165 that have a value at or above the cut-point were considered treatment-emergent ADA-positive. The number of participants with change from Baseline to any time post Baseline in the results of immunogenicity assessment as indicated by: negative to positive, positive to positive, positive to negative and negative to negative are presented.
Time Frame: Up to Week 22
Population: Intent-to-Treat Population. Only those participants with data available post-Baseline are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180mg
Number analyzed (Participants) | 22 | 22
Participants
  Negative to positive | 0 | 1
  Positive to positive | 0 | 0
  Positive to negative | 0 | 0
  Negative to negative | 22 | 20

17. Secondary Outcome: Apparent Clearance After Subcutaneous Administration (CL/F) of GSK3196165
Description: Blood samples were collected at indicated time points and CL/F was estimated using population PK analysis. Participants in the 'Safety' population who have at least one valid PK assessment were included Pharmacokinetic (PK) Population.
Time Frame: Day 3 and Pre-dose on Week 1, Week 4, Week 6, Week 12 and Week 22
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per day
Arm/Group | GSK3196165 180mg
Number analyzed (Participants) | 21
Liters per day | 4.94 (68.8)

18. Secondary Outcome: Apparent Steady State Volume of Distribution After Subcutaneous Administration (Vss/F) of GSK3196165
Description: Blood samples were collected at indicated time points and Vss/F was estimated using population PK analysis.
Time Frame: Day 3 and Pre-dose on Week 1, Week 4, Week 6, Week 12 and Week 22
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK3196165 180mg
Number analyzed (Participants) | 21
Liters | 36.5 (61.5)

19. Secondary Outcome: Absoption Rate Constant (Ka) of GSK3196165
Description: Blood samples were collected at indicated time points and Ka was estimated using population PK analysis.
Time Frame: Day 3 and Pre-dose on Week 1, Week 4, Week 6, Week 12 and Week 22
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per day
Arm/Group | GSK3196165 180mg
Number analyzed (Participants) | 21
Per day | 0.205 (72.3)

20. Secondary Outcome: Serum Concentration of GSK3196165 by Visit
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: Pre-dose on Day 3, Weeks 1, 4, 6, 12, follow up (Week 22)
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- GSK3196165 180 mg: Participants randomized to GSK3196165 group received total of 8 doses of GSK3196165 over a 12-week treatment period. Participants were administered loading doses on Days 1, 8, 15, 22 and 29 which was followed by 3 doses every other week (Days 43, 57, 71).
Arm/Group | GSK3196165 180 mg
Number analyzed (Participants) | 22
Nanogram per milliliter
  Day 3, n= 18: number analyzed (Participants) | 18
  Day 3, n= 18 | 2457.05 (94.74)
  Week 1, n= 21: number analyzed (Participants) | 21
  Week 1, n= 21 | 1767.55 (46.96)
  Week 4, n= 21: number analyzed (Participants) | 21
  Week 4, n= 21 | 2821.12 (61.00)
  Week 6, n= 20: number analyzed (Participants) | 20
  Week 6, n= 20 | 1802.09 (60.42)
  Week 12, n= 8: number analyzed (Participants) | 8
  Week 12, n= 8 | 800.96 (176.33)
  Follow up (Week 22), n= 12: number analyzed (Participants) | 12
  Follow up (Week 22), n= 12 | 56.40 (346.41)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) and serious AEs were collected up to Week 22.
Description: Non-serious AEs and SAE for Safety Population was reported.
Arm/Group | Placebo | GSK3196165 180mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/22
Other Adverse Events (participants affected / at risk) | 4/22 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | GSK3196165 180mg (N=22)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | GSK3196165 180mg (N=22)
PALPITATIONS (Cardiac disorders) | 2 (2) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 2 (3)
INJECTION SITE RASH (General disorders) | 0 (0) | 2 (6)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (3)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02683785/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT02683785/SAP_001.pdf